CLINICAL TRIAL: NCT04464213
Title: Phase I Clinical Trials of Human Placental Mesenchymal Stem Cells Treatment on Diabetic Foot Ulcer
Brief Title: Human Placental Mesenchymal Stem Cells Treatment on Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS201901
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Human placental mesenchymal stem cells; Gel
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose experiments (Experimental)
  Interventions: Other: Single dose experiments
- Multi-dose experiments (Experimental)
  Interventions: Other: Multi-dose experiments

INTERVENTIONS:
Other: Single dose experiments — In single dose experiments, after clean the diabetic foot ulcer, paint the Human placental mesenchymal stem cells gel on the wound, each patient only receive treatment once time.
  Arms: Single dose experiments
Other: Multi-dose experiments — In multi-dose experiments, after clean the diabetic foot ulcer, paint the Human placental mesenchymal stem cells gel on the wound, each patient receive treatment on six consecutive days.
  Arms: Multi-dose experiments

SUMMARY:
This study is designated to:

1. investigate the tolerance and safety of treatment of Human placental mesenchymal stem cells gel on Human diabetic foot ulcer.
2. learn the primary effectiveness of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.
3. study the pharmacokinetics of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and Age ≤ 75
* Type 1 or type 2 diabetes mellitus, glycosylated hemoglobin ≤ 9.0%
* Diagnosed as condition of diabetic foot ulcer, Wagner grade at 1 or 2 after clinical treatment
* Full understand the informed consent form, and signed it voluntarily

Exclusion Criteria:

* Pregnant or breast-feed women or plan to pregnant or fail to take an efficient contraception
* Be allergic to any component of the drug or showed allergic constitution
* Showed a sign of systemic infection, or with complication of ethmyphitis, or osteomyelitis indicated by MRI
* Have malignancy in the ulcer pathology test, or have a history of malignant tumor
* Unable to clean the wounds due to the formation of tract between the ulcer and other condition
* Infected with hepatitis B virus (HBV), hepatitis virus C (HCV), human immunodeficiency virus (HIV), or treponema pallidum
* Alanine transaminase (ALT) or aspartate transaminase (AST) exceeds 2.5 times of the normal value, or Cr>200 μmol/L
* Have a history of apoplexy, unstable angina pectoris, myocardial infarct
* Have a psychiatric history, drug abuse or alcohol abuse history
* Had participated in any other clinical trials in the past 3 months
* Any other circumstances judged by the researchers disqualify the patient to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse event | 0 hour - 24 hours
  The rate of adverse event in 24 hours after single dose of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.
Rate of adverse event | 0 Day - 7 Days
  The rate of adverse event in 7 days after multi-dose of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.

SECONDARY OUTCOMES:
Rate of serious adverse event | 0 hour - 1 hour
  The rate of serious adverse event in 1 hour after single dose of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.
Rate of cure rate | 0 day - 34 days
  Rate of cure rate in 20 days and 34 days after multi-dose of Human placental mesenchymal stem cells gel on Human diabetic food ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Doc, Principal Investigator — Beijing Tongren Hospital, CMU
Locations (1):
- National Institute for Drug Clinical Trial, Beijing Tongren Hospital, Capital Medical University, Beijing, Beiijng, China